CLINICAL TRIAL: NCT00834002
Title: Wilms Tumor Gene (WT1) mRNA-transfected Autologous Dendritic Cell Vaccination for Patients With Acute Myeloid Leukemia (AML): a Phase I Trial
Brief Title: Dendritic Cell Vaccination for Patients With Acute Myeloid Leukemia in Remission
Acronym: CCRG 05-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Prof dr Zwi Berneman, University Hospital Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC 5/6/29
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2009-08

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: AML in remission
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: injection of antigen-loaded cultured dendritic cells — intradermal injection of WT1-RNA-electroporated autologous dendritic cell vaccine (therapeutic cell vaccine)

SUMMARY:
RATIONALE: Vaccines made from a patient's white blood cells (dendritic cells) and a specific leukemia antigen (Wilms tumor antigen-1) may induce an effective immune response to kill residual leukemic cells and/or prevent leukemia relapse.

PURPOSE: This phase I/II trial is studying the feasibility, safety and efficacy of intradermal mRNA-transfected dendritic cell vaccination therapy in patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
Autologous dendritic cell (DC) vaccination is a promising strategy for adjuvant cancer therapy in the setting of minimal residual disease (MRD). We performed a phase I/II trial in patients with acute myeloid leukemia (AML) where patients received intradermal injections of autologous DC loaded with mRNA coding for the Wilms' tumor protein (WT1). WT1 is highly overexpressed in leukemia and the level of WT1 RNA in peripheral blood is a useful biomarker for molecular diagnosis en follow-up in the MRD setting. We want to prospectively monitor WT1 RNA expression in the peripheral blood of vaccinated and non-vaccinated AML patients in order to evaluate its predictive value as a biomarker for relapse and to assess the clinical efficacy of DC vaccination in acute myeloid leukemia patients. We believe, on the basis of already available evidence, that the use of WT1 both as a target for immunotherapy as well as a biomarker not holds promise to assess the efficacy of new experimental therapeutic interventions such as DC vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor type: Acute Myeloid Leukemia (AML) according to the WHO criteria (ea at least 20% blasts in the marrow). All FAB subtypes except M3. Patients with Myelodysplastic Syndrome, category of Refractory Anemia with Excess Blasts (RAEB): RAEB I (WHO: medullary blast count ≤ 10% and a peripheral blast count ≤ 5%) and RAEB II (WHO: medullary blast count > 10% and/or > 5% peripheral blasts) can be included in the study in absence of other non-experimental treatment modalities.
2. Extent of disease: remission (partial or complete) or smouldering course. Complete remission (CR) is defined as no blasts in the peripheral blood and no more than 5% blasts in the bone marrow. This definition is related to the hematological remission if it is not specified. Partial remission (PR) is defined as a decrease of at least 50% in the percentage of blasts to 5 to 25% in the bone marrow aspirate. Smouldering course is defined as a relatively low marrow blast count and slowly progressive disease.
3. Overexpression of WT1 RNA (>50 copies of WT1 per 1000 copies ABL in bone marrow or >2 copy/1000 copies ABL in peripheral blood) as assessed by quantitative RT-PCR at the time of presentation.
4. Prior treatments : Patients must have received at least one prior antileukemic chemotherapeutic regimen and must be more than 1 month past the last treatment and/or 6 months past allogeneic/autologous stem cell transplantation.
5. Age: ≥ 18 years
6. High risk of relapse because of (and/or)

   * Age > 60 years (if <60 y, no sibling allotransplant donor available)
   * Poor risk cytogenetic or molecular markers at presentation
   * Hyperleukocytosis at presentation
   * Second complete remission after relapse
7. Performance status: WHO PS grade 0-1 (Appendix B)
8. Objectively assessable parameters of life expectancy: more than 3 months
9. Prior and concomitant associated diseases allowed with the exception of underlying autoimmune disease and positive serology for HIV/HBV/HCV
10. No concomitant use of immunosuppressive drugs
11. Adequate renal and liver function, i.e. creatinin and bilirubin = 1.2 times the upper limit of normal
12. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
13. Women of child-bearing potential should use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

1. Subjects with concurrent additional malignancy (with exception of Non-melanoma skin cancers and carcinoma in situ of the cervix)
2. Subjects who are pregnant
3. Subjects who have sensitivity to drugs that provide local anesthesia
4. Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-03; Primary Completion 2007-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
acute toxicity of intradermal injections of WT1 mRNA-electroporated autologous dendritic cells
feasibility to generate functional DC vaccines from leukapheresis material from AML patient in remission

SECONDARY OUTCOMES:
T cell immunogenicity of WT1 mRNA-loaded dendritic cell vaccines in AML patients in remission

CONTACTS AND LOCATIONS:
Overall Officials: Zwi Berneman, MD, PHD, Study Director — University Hospital, Antwerp; Ann Van de Velde, MD, Principal Investigator — University Hospital, Antwerp; Viggo FI Van Tendeloo, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital/Center for Cellular Therapy and Regenerative Medicine, Edegem, Belgium